CLINICAL TRIAL: NCT02778802
Title: Pulmonary Hemodynamics in Patients With Severe Emphysema Pre and Post Bronchoscopic Volume Reduction by Histoacryl or Silver Nitrate (Single Center Experince )
Brief Title: Pulmonary Hemodynamics in Patients With Severe Emphysema Pre and Post BLVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Elshazly, Professor of pulmonary Medicine, Cairo University
Other Study IDs: Cairo2002
Record Dates: First submitted 2016-05-14; First posted 2016-05-20 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Lung Disease
Keywords: Pulmonary Hypertension; Emphysema; COPD
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed as a prospective study, with the primary endpoint being changes in pulmonary hemodynamic parameters after ELVR in patients with severe emphysema.

Secondary endpoints will be changes in lung function parameters, exercise capacity, and QoL.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) continues to be a leading cause of morbidity and is currently the third most common cause of mortality worldwide (1).

In most patients with severe COPD, chronic airflow limitation, lung emphysema with parenchymal destruction and the development of air bullae also occur (2-3) Pulmonary hypertension (PH) is a common consequence of COPD, although the actual overall prevalence of PH in COPD remains unclear (4). Among COPD patients who were to undergo lung-volume-reduction surgery or lung transplantation, mild PH was observed in 50.2%, moderate PH in 9.8%, and severe PH in 3.7%(5). While in most COPD patients who develop PH, pulmonary arterial pressure is only mildly or moderately elevated, (6) PH has an independent prognostic impact on survival. (6,7) The therapeutic options for COPD patients with severe emphysema are limited. Lung volume reduction surgery (LVRS) has been performed as treatment in selected cases, but the referral of patients has been severely influenced by the marked perioperative morbidity and mortality [8]. Less invasive techniques have been developed with the aim of improving patients' pulmonary function, symptoms, and quality of life (QoL) [9]. Among them, the one most commonly used is the endoscopic placement of one way endobronchial valves (EBV) [10-12]. So far patients with severe emphysema and established PH have been excluded from LVRS as well as from endoscopic lung volume reduction (ELVR) therapy.

Whether bronchoscopic lung volume reduction in COPD patients with silver nitrate or histoacryl influences the severity of PH in patients with severe emphysema and PH has yet to be elucidated.

This study is designed as a prospective pilot study, with the primary endpoint being changes in pulmonary hemodynamic parameters after ELVR in patients with severe emphysema.

Secondary endpoints will be changes in lung function parameters, exercise capacity, and QoL.

Materials and Methods This is Prospective descriptive study on 20 COPD Patients with predominant emphysema especially with heterogeneous and upper lobe predominance emphysema admitted in chest department at Kasr al Ainy Hospital. All patients will be on optimal medical treatment for COPD according to Global Initiative for Chronic Obstructive Lung Disease guidelines [13] All patients will be subjected to the following at base line.

1. full history taking.
2. full clinical examination.
3. plain chest x ray.
4. an electrocardiogram, High resolution computed tomography of the chest.
5. Pulmonary function tests and ABG.
6. 6-minute walk test.
7. 2-D echocardiography at rest
8. Right heart catheterization (RHC)
9. Fiberoptic bronchoscopy with application of silver nitrate or histoacryl. The patients will be followed up every month by

1. Dyspnea score (using mMRC score) 2. 6-minute walk test. 3. ECG At 3rd Month 2-D echocardiography at rest will be done At 6th Month 2-D echocardiography at rest And RHC will be done .

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with predominant emphysema especially with heterogeneous and upper lobe predominance emphysema

Exclusion Criteria:

1. Airflow limitation with FEV1 < 20%.
2. Patients not candidate for FOB.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD Patients with predominant emphysema especially with heterogeneous and upper lobe predominance emphysema
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
change in mean Pulmonary artery pressure after ELVR | 3months, 6monthes
  Right heart cathetrization

SECONDARY OUTCOMES:
Dysnea Score | 3 months,6months
  using modified Medical Research Council (mMRC) criteria, with 0 representing dyspnea with strenuous exercise and 4 representing dyspnea with breathlessness when dressing

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elnady, MD, Study Director — Professor of pulmonary Medicine ,Cairo University; Karim Mahmoud, MD, Study Director — Lecturer of cardiology ,Cairo University
Locations (1):
- Kasr Alaini School of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer reviewed Journal